CLINICAL TRIAL: NCT06679023
Title: Biofilms in Chronic Wounds Pathogenesis and Diagnosis: Quantification of Biofilm and Validation of Grading System in Modified Alcian Blue Biofilm Detection Kit (WBDK-GB)
Brief Title: Wound Biofilm Detection Kit Development: Validation of Grading System With Biofilm Severity
Acronym: WBDK-GB
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202304083DINB
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: Chronic Wound; Wound Healing; Biofilm Infection
Keywords: chronic wound; wound healing; Biofilm detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — chronic wound specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MolecuLight i:X and Wound blotting and Alcian blue biofilm detection kit — we will enroll patients with chronic wounds and quantify the biofilm severity by staining color of Wound blotting and Alcian blue biofilm detection kit, and by non-touched flourescent intensity of MolecuLight i:X.

SUMMARY:
Chronic wound is a leading health issue in current health care system. Biofilm is a notorious risk factor of unhealed wound. Although biofilm-direct wound care has been a prevalent strategy of wound care currently, diagnosis of biofilm still remained as an unmet clinical need. Several advanced diagnostic tools of biofilm had been published in recent years, however, the evidence was still insufficient.

In this study, we will enroll patients with chronic wounds, collect the wound debris, quantify the biofilm and validate with the signals of advanced diagnostic tools for biofilm detection, hoping to transform the tools which could only tell us whether the biofilm is present or not, into the severity of biofilm infection. The two tested tools includes of MolecuLight i:X and wound blotting and Alcian blue biofilm detection kit.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18 or older
* 2.Has an unhealed wound and is scheduled for debridement surgery
* 3.Patients who are receiving wound care at this hospital (Hsinchu branch) and are able to comply with follow-up wound monitoring

Exclusion Criteria:

* Does not consent to provide remaining tissue from wound treatment for in vitro analysis.
* Allergic to nylon components.
* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic wound
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
90-day wound healing | 90 days
  observation 90-day wound healing and its relationship with clinical data and biofilm severity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No